CLINICAL TRIAL: NCT00423748
Title: Ambrisentan in PAH - A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Efficacy Study of Ambrisentan in Subjects With Pulmonary Arterial Hypertension
Brief Title: Study to Assess Safety and Efficacy of Ambrisentan in Subjects With Pulmonary Arterial Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMB-320; ARIES-1
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2009-04-16 (Estimated); Status verified 2009-04

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

INTERVENTIONS:
Drug: ambrisentan

SUMMARY:
A phase 3, randomized, double-blind, placebo-controlled study to assess safety and efficacy of ambrisentan in subjects with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Subjects in these randomized studies will receive one of two doses of ambrisentan or placebo. Inclusion is not based on a specified WHO functional classification. Rather, subjects with WHO Class I-IV symptoms are eligible if their 6-minute walk distance is 150-450 meters and they meet the study-specified hemodynamic criteria. Subjects with anorexigen or HIV infection related PAH are eligible but subjects with congenital heart disease and pediatric subjects are excluded. The study requires a historical cardiac catheterization and other diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or order
* Current diagnosis of either PPH orPAH secondary to the scleroderma spectrum of disease, systemic lupus erythematosus, anorexigen use, or HIV infection at the Screening Visit
* Right heart catheterization, completed prior to Screening Visit must meet pre-specified hemodynamic criteria
* Female subjects of childbearing potential must have a negative serum pregnancy test and must agree to use a reliable double barrier method of contraception until study completion and for at least four weeks following their final study visit
* Male subjects must be informed of the potential risks of testicular tubular atrophy and infertility associated with taking this study drug and queried regarding his understanding of the potential risks as described in the Informed Consent Form

Exclusion Criteria:

* PAH due to or associated with congenital heart disease, coronary artery disease, left heart disease, interstitial lung disease, chronic obstructive pulmonary disease, veno-occlusive disease, chronic thrombotic and/or embolic disease, or sleep apnea
* Portopulmonary hypertension
* Bosentan within four weeks prior to Screening
* Phosphodiesterase type V inhibitor or chronic prostanoid therapy within four weeks prior to Screening
* IV inotrope use within two weeks prior to Screening
* ALT or AST lab value that is greater than 1.5 times the upper limit of normal
* Pulmonary function tests not meeting pre-specified criteria
* Contraindication to treatment with an ERA
* History of malignancies other than basal cell carcinoma of the skin or in situ carcinoma of the cervix within the past five years
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2003-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Change from baseline in the six-minute walk distance evaluated after 12 weeks of therapy compared to placebo.

SECONDARY OUTCOMES:
Change from baseline measured after 12 weeks of treatment compared to placebo in the Borg Dyspnea Index; WHO Functional Classification; and the SF-36 Health Survey.
Clinical worsening of PAH.
Assessment of the safety and tolerability of the study drug.